CLINICAL TRIAL: NCT07050121
Title: A Prospective Multi-Center Real-World Study of Ciwujia Capsules in the Treatment of Cancer-Related Insomnia
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Municipal Hospital of Traditional Chinese Medicine (Other)
Collaborators: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Henan Provincial Hospital of Integrated Traditional Chinese and Western Medicine (Unknown); Shanghai East Hospital (Other); Bao'an Authentic TCM therapy Hospital (Unknown); Chengdu Fifth People's Hospital (Other); Chengdu Shuangliu Traditional Chinese Medicine Hospital (Unknown); Ezhou Traditional Chinese Medicine Hospital (Unknown); Shanghai 7th People's Hospital (Other); The Affiliated Hospital of Shaanxi University of Traditional Chinese Medicine (Unknown); Putuo District Central Hospital of Shanghai (Unknown); Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025SHSZYYYRWS
Record Dates: First submitted 2025-06-12; First posted 2025-07-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Insomnia; Cancer Related Insomnia
MeSH Terms: conditions — Neoplasms; Sleep Initiation and Maintenance Disorders | interventions — Siberian ginseng root

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 56 Days
Biospecimen Retention: Samples Without DNA — This study collects blood and urine samples from participants for safety assessments; however, sample collection is not mandatory and will be conducted solely based on participants' voluntary consent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Naturally Exposed Group: Patients voluntarily taking Ciwujia capsules, Ciwujia capsules for oral use，2-3 capsules per dose, three times daily. 28 days constitute one treatment course; efficacy and safety will be assessed over two courses. Dosage adjustments should follow the physician's instructions.
  Interventions: Drug: Ciwujia capsules

INTERVENTIONS:
Drug: Ciwujia capsules — Ciwujia capsules for oral use，2-3 capsules per dose, three times daily. 28 days constitute one treatment course; efficacy and safety will be assessed over two courses. Dosage adjustments should follow the physician's instructions.

SUMMARY:
Cancer poses a severe threat to human physical and mental health as well as survival. High diagnostic rates of cancer and various treatments can significantly impact patients' sleep quality, leading to diverse sleep disorders. Cancer-related insomnia (CRI) is a prevalent sleep disturbance among cancer patients, potentially associated with the tumor itself, treatment modalities (such as surgery, chemotherapy, radiotherapy), psychological status, pain, fatigue, and other symptoms. Although reported incidence rates vary across studies, CRI is consistently high and severely compromises patients' quality of life. Core symptoms include difficulty falling asleep, sleep maintenance difficulties, and early morning awakening, which contribute to daytime fatigue, impaired concentration and memory, ultimately detrimentally affecting patients' health and quality of life. The pathogenesis of CRI is complex, potentially involving multiple factors including the tumor's direct effects, treatment side effects, psychological distress, pain, and fatigue.

The primary component of Ciwujia capsules (containing Eleutherococcus senticosus extract) is Ciwujia extract. To clarify the clinical efficacy of Ciwujia capsules for cancer-related insomnia in real-world clinical settings, this study will employ a multicenter, prospective, open-label, real-world research design. It is projected to involve 30-50 centers over an approximate 3-year trial period, with a planned enrollment of 3,000 subjects. Changes in sleep-related indicators before and after treatment will serve as the primary endpoint observation metrics. The study aims to investigate the clinical efficacy and safety profile of Ciwujia capsules in treating insomnia disorders in cancer patients, thereby providing robust evidence for identifying effective Chinese herbal medicine therapies for sedation and sleep promotion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤75 years.
2. Histologically and/or cytologically confirmed diagnosis of malignancy. 3.Meet the diagnostic criteria for insomnia disorder per the Chinese Guidelines for Diagnosis and Treatment of Insomnia in Adults (2023) with one of the following conditions: 1）Directly cancer-related insomnia: Insomnia symptoms (e.g. difficulty falling asleep sleep maintenance difficulties early awakening) directly attributable to cancer-associated factors: ① Tumor-related factors: Pain cachexia dyspnea cough pruritus tumor compression symptoms etc. ② Cancer treatment-related factors: Chemotherapy-induced nausea/vomiting post-radiation mucositis surgical trauma etc. ③ Cancer-associated complications: Anemia infections metabolic disturbances etc. 2）Indirectly cancer-related insomnia: Insomnia directly caused by psychological stress reactions to cancer diagnosis or disease progression such as fear/anxiety about disease progression concerns about treatment side effects financial burden or psychosocial factors (e.g. insufficient family support).

4.Eastern Cooperative Oncology Group (ECOG) performance status score of 0-3. 5.Voluntarily participate and provide written informed consent.

Exclusion Criteria:

1. History of allergy to any component of the investigational product.
2. Liver dysfunction with ALT/AST levels exceeding 1.5 times the upper limit of normal (ULN).
3. Severe psychiatric disorders or emotional disturbances within the past year (e.g. anxiety depression suicidal tendencies or suicide attempts) requiring long-term use of CNS depressants or stimulants.
4. Women who are pregnant breastfeeding or of childbearing potential unwilling to use effective contraception during the study.
5. Insomnia secondary to uncontrolled severe cancer-related pain. 6.Participation in another clinical drug trial within the past month.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The purpose of this study is to evaluate the efficacy and safety of Ciwuja capsules in treating cancer-related insomnia in a real-world clinical setting. Cancer patients eligible for participation are not restricted by cancer type, disease stage, or treatment regimen, and may be enrolled after meeting the study's inclusion and exclusion criteria screening.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Assessments at baseline，day28±5，day56±5

SECONDARY OUTCOMES:
Individual Components of the Pittsburgh Sleep Quality Index (PSQI) | Assessments at baseline，day28±5，day56±5
  Including sleep latency, subjective sleep quality, sleep continuity, habitual sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction. Each component will be assessed.
Insomnia Severity Index (ISI) | Assessments at baseline，day14±3，day28±5，day56±5
EORTC QLQ-C30 | Assessments at baseline，day14±3，day28±5，day56±5

OTHER OUTCOMES:
Pharmacoeconomic Evaluation | Assessments were performed after day 56 post-enrollment.
  Conduct a pharmacoeconomic cost-effectiveness analysis, the unit cost of effectiveness is calculated by dividing the total drug-related expenses incurred during treatment - comprising direct costs (medication expenses) plus indirect costs (such as registration, transportation fees and so on) - by the change in PSQI scores before versus after drug administration.
Alanine Aminotransferase(ALT) | Assessments at baseline, day56±5
  Non-mandatory indicators, tested based on patient preference
Urine Protein | Assessments at baseline, day56±5
  Non-mandatory indicators, tested based on patient preference
White Blood Cell | Assessments at baseline, day56±5
  Non-mandatory indicators, tested based on patient preference
Aspartate Aminotransferase(AST) | Assessments at baseline, day56±5
  Non-mandatory indicators, tested based on patient preference
Serum Creatinine | Assessments at baseline, day56±5
  Non-mandatory indicators, tested based on patient preference
Urine Occult Blood | Assessments at baseline, day56±5
  Non-mandatory indicators, tested based on patient preference
Hemoglobin | Assessments at baseline, day56±5
  Non-mandatory indicators, tested based on patient preference
Platelet | Assessments at baseline, day56±5
  Non-mandatory indicators, tested based on patient preference
Electrocardiogram QT Interval | Assessments at baseline, day56±5
  Non-mandatory indicators, tested based on patient preference

CONTACTS AND LOCATIONS:
Overall Officials: Jianhui Tian, Doctor, Study Director — Shanghai Municipal Hospital of Traditional Chinese Medicine - Oncology Research Center

IPD SHARING:
Plan to Share IPD: Undecided